CLINICAL TRIAL: NCT01575171
Title: Using Nudges to Implement Comparative Effectiveness: Behavioral Economics and Statins
Brief Title: Using Nudges to Implement Comparative Effectiveness
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 10-01287
Record Dates: First submitted 2012-04-02; First posted 2012-04-11 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Intervention/"Nudge": Individuals will be analyzed according to their assigned intervention group, to compare the effectiveness of an opt-out EHR decision support system to enhance the prescription of statins to those patients with an elevated LDL-C and to subsequently titrate the medication dose until LDL-C control is obtained. Physicians randomized to the automated clinical decision support "nudge" will see the new "optout" prescribing procedure as part of their EHR interface. This will include initially prescribing the guideline-based medication, simvastatin 20mg. Nearly six months after this visit, physicians will receive a reminder via EHR to schedule a follow-up fasting lipid profile as recommended by ATP III guidelines.
  Interventions: Behavioral: Nudge

INTERVENTIONS:
Behavioral: Nudge — Behavioral economics recognizes that individuals often are not fully "rational" in the purely economic sense, but are subject to the influence of various social, environmental and cognitive factors in their decision making. And, one can take advantage of these findings to "nudge" individuals, in our case physicians, towards more optimal choices. Physicians randomized to the automated clinical decision support "nudge" will see the new "optout" prescribing procedure as part of their EHR interface. This will include initially prescribing the guideline-based medication, simvastatin 20mg. Nearly six months after this visit, physicians will receive a reminder via EHR to schedule a follow-up fasting lipid profile as recommended by ATP III guidelines.

SUMMARY:
Behavioral economics represents a powerful, albeit underutilized tool to influence provider and systems behavior in a large-scale, meaningful, and sustainable way. The investigators propose to use a sophisticated electronic health record (EHR) system to change the default choice for physicians to the choice most supported by clinical practice guidelines (CPG).

Multiple guidelines exist describing best practices for effective interventions, yet a large gap persists between actual and optimal guideline compliance. The proposed study will examine the comparative effectiveness of an opt-out medication management protocol relative to usual care for patients not at goal, using national guidelines for cholesterol management implemented in large multispecialty private practices that use an Electronic Health Record system.

Specific Aim: To determine the effectiveness of altering the default option in an EHR in prescribing statins to selected patients using clinical decision support.

Hypotheses: Compared to usual care, a CPG-concordant intervention designed using behavioral economics principles will significantly improve the proportion of patients who are prescribed statins.

DETAILED DESCRIPTION:
Historically, many interventions have been studied to improve the quality, safety, and effectiveness of medical care, particularly through the new focus on comparative effectiveness research. Unfortunately, sustained provider and system uptake of these interventions has been severely lacking, to the serious detriment of patient health. The most commonly tried tools to increase uptake, including pay-for-performance, have substantially fallen short of expectations. Moreover, often these interventions are created in highly artificial settings, and we have not come up with ways to implement them in the long-term. The challenge, therefore, is to create sustainable change that impacts care in meaningful ways.

In contrast, behavioral economics represents a powerful tool by which to influence provider and systems behavior in a large-scale, meaningful, and sustainable way. Briefly, behavioral economics recognizes that individuals often are not fully "rational" in the purely economic sense, but are subject to the influence of various social, environmental and cognitive factors in their decision making. And, one can take advantage of these findings to "nudge" individuals, in our case physicians, towards more optimal choices. While the application of behavioral economics has been incredibly successful in altering behavior outside the health sphere, surprisingly little attention has been given to health.

We have chosen to focus on physician behavior in prescribing HMG-CoA reductase inhibitors (statins) to patients with elevated cardiac risk and elevated low density lipoprotein cholesterol (LDL-C) as recommended by cholesterol management guidelines. In a cluster randomized trial at several private, community-based, multispecialty practices, we propose to compare usual care to a system of automated, default, opt-out clinical decision support that prescribes statins as appropriate.

We propose to use a cluster randomized trial design in several multispecialty private practices to examine the comparative effectiveness of an EHR-based lipid management protocol based on ATP III guidelines vs. usual care. Cluster randomization of participating physicians is useful when blinding is impossible and "contamination" might be a problem, i.e. more aggressive management among a physician's non-intervention patients as a result of experience with intervention patients. Of an estimated 150 primary care physicians at the recruited private practices, we expect at least 100 to consent to participate. Physicians will be clustered for randomization based on the number of patients in their panel that meet ATP III guidelines for statin. Physicians in each cluster will then be individually randomized to the intervention or control arm.

Physicians randomized to usual care will not get the intervention or decision support. Physicians randomized to the automated clinical decision support "nudge" will see the new "optout" prescribing procedure as part of their EHR interface. This will include initially prescribing the guideline-based medication, simvastatin 20mg. Nearly six months after this visit, physicians will receive a reminder via EHR to schedule a follow-up fasting lipid profile as recommended by ATP III guidelines.

ELIGIBILITY:
Doctors who have patients that meet the inclusion/exclusion criteria below.

Inclusion Criteria:

* Male patients 18+
* Female patients age 50+ (to avoid the possibility of women of childbearing age being started on statin)
* Fasting lipid profile from the past year who meet ATP III guidelines for requiring a statin

Exclusion Criteria:

* Women less than 50 years of age
* Patients with allergy/myopathy to statins in the past
* Patients with active liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Doctors in a large multi-specialty private practice
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2010-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Nudge Acceptance or Rejection | Doctor visit to 6 months
  A "Nudge" or opt-out default option is implemented in the electronic health record system based on national clinical guidelines. We plan to measure if the Nudge is accepted or rejected by doctors.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ravenell, MD, MS, Principal Investigator — NYU School of Medicine; Brian Elbel, PhD, MPH, Principal Investigator — NYU School of Medicine
Locations (1):
- Murray Hill Medical Group, New York, New York, United States